CLINICAL TRIAL: NCT05767710
Title: An Alternative Remote Rehabilitation Strategy for the Improvement of Sarcopenia in the Elderly: Tai Chi as an Exercise Form
Brief Title: A Study of the Telerehabiliation Intervention Effect of the Tai Chi Exercise on Elderly With Sarcopenia
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Northeast Normal University (Other)
Responsible Party: Principal Investigator, Guang Yang, Prof. Dr., Prof.Dr., Northeast Normal University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: CCEE2023
Record Dates: First submitted 2023-03-02; First posted 2023-03-14 (Actual); Last update posted 2023-03-14 (Actual); Status verified 2023-03

CONDITIONS: Sarcopenia
Keywords: sarcopenia; human pose
MeSH Terms: conditions — Sarcopenia

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (9):
- AI telerehabilitation - Tai Chi (Experimental): All sessions were conducted online, with participants practicing along with Tai Chi videos while the AI guided the movements throughout the session. A remote rehabilitation program was installed in patients' homes by study team members. Participants who do not know how to use a computer were assisted by their family members.
  Interventions: Behavioral: AI telerehabilitation - Tai Chi
- general telerehabilitation - Tai Chi (Active Comparator): All sessions were conducted in an online format, with participants practicing along with Tai Chi videos while the professional Tai Chi instructors supervised and guided the movements throughout the session. A computer connected to a high-resolution webcam was used to establish real-time remote visual communication between the rehabilitation unit and the patient's home via Tencent conferencing software (Meeting/Tencent).
  Interventions: Behavioral: general telerehabilitation - Tai Chi
- traditional rehabilitation - Tai Chi (Active Comparator): All sessions were conducted offline and implemented by professional Tai Chi instructors. The audio from the video used for the other two groups was utilized to assist the practice of participants in traditional rehabilitation - Tai Chi group.
  Interventions: Behavioral: traditional rehabilitation - Tai Chi
- AI telerehabilitation - Yi Jin Jing (Experimental): All sessions were conducted online, with participants practicing along with Yi Jin Jing videos while the AI guided the movements throughout the session. A remote rehabilitation program was installed in patients' homes by study team members. Participants who do not know how to use a computer were assisted by their family members.
  Interventions: Behavioral: AI telerehabilitation - Yi Jin Jing
- general telerehabilitation - Yi Jin Jing (Active Comparator): All sessions were conducted in an online format, with participants practicing along with Yi Jin Jing videos while the professional Yi Jin Jing instructors supervised and guided the movements throughout the session. A computer connected to a high-resolution webcam was used to establish real-time remote visual communication between the rehabilitation unit and the patient's home via Tencent conferencing software (Meeting/Tencent).
  Interventions: Behavioral: general telerehabilitation - Yi Jin Jing
- traditional rehabilitation - Yi Jin Jing (Active Comparator): All sessions were conducted offline and implemented by professional Yi Jin Jing instructors. The audio from the video used for the other two groups was utilized to assist the practice of participants in traditional rehabilitation - Yi Jin Jing group.
  Interventions: Behavioral: traditional rehabilitation - Yi Jin Jing
- AI telerehabilitation - Ba Duan Jin (Experimental): All sessions were conducted online, with participants practicing along with Ba Duan Jin videos while the AI guided the movements throughout the session. A remote rehabilitation program was installed in patients' homes by study team members. Participants who do not know how to use a computer were assisted by their family members.
  Interventions: Behavioral: AI telerehabilitation - Ba Duan Jin
- general telerehabilitation - Ba Duan Jin (Active Comparator): All sessions were conducted in an online format, with participants practicing along with Ba Duan Jin videos while the professional Ba Duan Jin instructors supervised and guided the movements throughout the session. A computer connected to a high-resolution webcam was used to establish real-time remote visual communication between the rehabilitation unit and the patient's home via Tencent conferencing software (Meeting/Tencent).
  Interventions: Behavioral: general telerehabilitation - Ba Duan Jin
- traditional rehabilitation - Ba Duan Jin (Active Comparator): All sessions were conducted offline and implemented by professional Ba Duan Jin instructors. The audio from the video used for the other two groups was utilized to assist the practice of participants in traditional rehabilitation - Ba Duan Jin group.
  Interventions: Behavioral: traditional rehabilitation - Ba Duan Jin

INTERVENTIONS:
Behavioral: AI telerehabilitation - Tai Chi — All the participants received a three-month intervention which consisted two stage: the first month was the movement learning and consolidation phase, with 45 minutes of Tai Chi practice per session and three times each week; the last two months were the formal practice phase with 45 minutes of Tai Chi practice per session and three times each week. In the first phase, participants learned four new movements in each session and consolidated these exercises in the next session. After all the movements have been learned, use the remaining time in the first stage to consolidate the exercises. In the second phase, participants performed a complete Tai Chi exercise in each session.
  Arms: AI telerehabilitation - Tai Chi
Behavioral: general telerehabilitation - Tai Chi — All the participants received a three-month intervention which consisted two stage: the first month was the movement learning and consolidation phase, with 45 minutes of Tai Chi practice per session and three times each week; the last two months were the formal practice phase with 45 minutes of Tai Chi practice per session and three times each week. In the first phase, participants learned four new movements in each session and consolidated these exercises in the next session. After all the movements have been learned, use the remaining time in the first stage to consolidate the exercises. In the second phase, participants performed a complete Tai Chi exercise in each session.
  Arms: general telerehabilitation - Tai Chi
Behavioral: traditional rehabilitation - Tai Chi — All the participants received a three-month intervention which consisted two stage: the first month was the movement learning and consolidation phase, with 45 minutes of Tai Chi practice per session and three times each week; the last two months were the formal practice phase with 45 minutes of Tai Chi practice per session and three times each week. In the first phase, participants learned four new movements in each session and consolidated these exercises in the next session. After all the movements have been learned, use the remaining time in the first stage to consolidate the exercises. In the second phase, participants performed a complete Tai Chi exercise in each session.
  Arms: traditional rehabilitation - Tai Chi
Behavioral: AI telerehabilitation - Yi Jin Jing — All the participants received a three-month intervention which consisted two stage: the first month was the movement learning and consolidation phase, with 45 minutes of Yi Jin Jing practice per session and three times each week; the last two months were the formal practice phase with 45 minutes of Yi Jin Jing practice per session and three times each week. In the first phase, participants learned four new movements in each session and consolidated these exercises in the next session. After all the movements have been learned, use the remaining time in the first stage to consolidate the exercises. In the second phase, participants performed a complete Yi Jin Jing exercise in each session.
  Arms: AI telerehabilitation - Yi Jin Jing
Behavioral: general telerehabilitation - Yi Jin Jing — All the participants received a three-month intervention which consisted two stage: the first month was the movement learning and consolidation phase, with 45 minutes of Yi Jin Jing practice per session and three times each week; the last two months were the formal practice phase with 45 minutes of Yi Jin Jing practice per session and three times each week. In the first phase, participants learned four new movements in each session and consolidated these exercises in the next session. After all the movements have been learned, use the remaining time in the first stage to consolidate the exercises. In the second phase, participants performed a complete Yi Jin Jing exercise in each session.
  Arms: general telerehabilitation - Yi Jin Jing
Behavioral: traditional rehabilitation - Yi Jin Jing — All the participants received a three-month intervention which consisted two stage: the first month was the movement learning and consolidation phase, with 45 minutes of Yi Jin Jing practice per session and three times each week; the last two months were the formal practice phase with 45 minutes of Yi Jin Jing practice per session and three times each week. In the first phase, participants learned four new movements in each session and consolidated these exercises in the next session. After all the movements have been learned, use the remaining time in the first stage to consolidate the exercises. In the second phase, participants performed a complete Yi Jin Jing exercise in each session.
  Arms: traditional rehabilitation - Yi Jin Jing
Behavioral: AI telerehabilitation - Ba Duan Jin — All the participants received a three-month intervention which consisted two stage: the first month was the movement learning and consolidation phase, with 45 minutes of Ba Duan Jin practice per session and three times each week; the last two months were the formal practice phase with 45 minutes of Ba Duan Jin practice per session and three times each week. In the first phase, participants learned four new movements in each session and consolidated these exercises in the next session. After all the movements have been learned, use the remaining time in the first stage to consolidate the exercises. In the second phase, participants performed a complete Ba Duan Jin exercise in each session.
  Arms: AI telerehabilitation - Ba Duan Jin
Behavioral: general telerehabilitation - Ba Duan Jin — All the participants received a three-month intervention which consisted two stage: the first month was the movement learning and consolidation phase, with 45 minutes of Ba Duan Jin practice per session and three times each week; the last two months were the formal practice phase with 45 minutes of Ba Duan Jin practice per session and three times each week. In the first phase, participants learned four new movements in each session and consolidated these exercises in the next session. After all the movements have been learned, use the remaining time in the first stage to consolidate the exercises. In the second phase, participants performed a complete Ba Duan Jin exercise in each session.
  Arms: general telerehabilitation - Ba Duan Jin
Behavioral: traditional rehabilitation - Ba Duan Jin — All the participants received a three-month intervention which consisted two stage: the first month was the movement learning and consolidation phase, with 45 minutes of Ba Duan Jin practice per session and three times each week; the last two months were the formal practice phase with 45 minutes of Ba Duan Jin practice per session and three times each week. In the first phase, participants learned four new movements in each session and consolidated these exercises in the next session. After all the movements have been learned, use the remaining time in the first stage to consolidate the exercises. In the second phase, participants performed a complete Ba Duan Jin exercise in each session.
  Arms: traditional rehabilitation - Ba Duan Jin

SUMMARY:
Sarcopenia is an age-related disease characterized by a progressive decrease in skeletal muscle content and loss of muscle function. Tai Chi exercises have been shown to improve skeletal muscle mass in elderly people suffering from sarcopenia. However, offline interventions are a very labor- and financial-intensive approach. Therefore, researchers designed an artificial intelligence-assisted program and Tai Chi exercise format to investigate whether a remote rehabilitation approach could replace face-to-face interventions

ELIGIBILITY:
Inclusion Criteria:

(1) Patients between the ages of 60-75 years; (2) who meet the screening criteria for sarcopenia in Asia established by AWGS 2019; (3) who have a computer at home (4) who can use a computer or was accompanied by family number who can use a computer.

Exclusion Criteria:

(1) participants taking medications that significantly impact musculoskeletal function (2) participants suffering from respiratory failure or other bodily problems; (3) participants with mental disorders or neurological disorders; (4) patients who participate in other training programs on a regular basis.

Ages: 60 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 225 (Estimated)
Dates: Start 2023-04-10 (Estimated); Primary Completion 2023-07-10 (Estimated); Study Completion 2023-07-20 (Estimated)

PRIMARY OUTCOMES:
Using quantitative CT to investigate the change of skeletal muscle area in sarcopenic elderly. | Month 3
  articipants will receive quantitative CT scans before and after the intervention to assess the change from baseline skeletal muscle area at 3 months.
Using a Jamar hydraulic hand dynamometer to investigate change of handgrip in sarcopenic elderly. | Month 3
  Participants will receive a handgrip strength test before and after the intervention to assess the change from baseline handgrip strength at 3 months.
Using a bioelectrical impedance body composition analyzer with a multifrequency device to investigate the change of relative skeletal muscle mass index in sarcopenic elderly. | Month 3
  Participants will receive a relative skeletal muscle mass index test before and after the intervention to assess the change from baseline relative skeletal muscle index at 3 months.

SECONDARY OUTCOMES:
Collect participants' self-evaluation of their life state and physical state. | Month 3
  Participants were asked to write a self-assessment report of no more than 500 words before and after the intervention, including physical status and life status.
Collect video of participants throughout the intervention. | Month 3
  The entire intervention process was recorded and video of the entire intervention process was collected from the participants.

CONTACTS AND LOCATIONS:
Locations (1):
- Chinese Center of Exercise Epidemiology, Changchun, Jilin, China

REFERENCES:
- [Derived] He S, Meng D, Wei M, Guo H, Yang G, Wang Z. Proposal and validation of a new approach in tele-rehabilitation with 3D human posture estimation: a randomized controlled trial in older individuals with sarcopenia. BMC Geriatr. 2024 Jul 8;24(1):586. doi: 10.1186/s12877-024-05188-7. PMID 38977995